CLINICAL TRIAL: NCT04802161
Title: Randomized Phase 2 Study of Daunorubicin and Cytarabine Liposome + Pomalidomide Versus Daunorubicin and Cytarabine Liposome in Newly Diagnosed AML With MDS-Related Changes
Brief Title: Comparing the Addition of an Anti-Cancer Drug, Pomalidomide, to the Usual Chemotherapy Treatment (Daunorubicin and Cytarabine Liposome) in Newly Diagnosed Acute Myeloid Leukemia With Myelodysplastic Syndrome-Related Changes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-01961; NCI-2021-01961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10434 (Other: Ohio State University Comprehensive Cancer Center LAO); 10434 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2021-03-16; First posted 2021-03-17 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Post Cytotoxic Therapy; Acute Myeloid Leukemia With Multilineage Dysplasia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Specimen Handling; Biopsy; CPX-351; Cytarabine; Daunorubicin; Injections; Liposomes; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (daunorubicin and cytarabine liposome, pomalidomide) (Experimental): INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 and then pomalidomide PO QD beginning between days 21-30 for 14 days in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Drug: Pomalidomide
- Arm B (daunorubicin and cytarabine liposome) (Active Comparator): INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspirate and biopsy
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX 351; CPX-351; CPX351; Cytarabine and Daunorubicin Liposomal; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC 4047; CC-4047; CC4047; Imnovid; Pomalyst
  Arms: Arm A (daunorubicin and cytarabine liposome, pomalidomide)

SUMMARY:
This phase II trial studies the effect of adding pomalidomide to usual chemotherapy treatment (daunorubicin and cytarabine liposome) in treating patients with newly diagnosed acute leukemia with myelodysplastic syndrome-related changes. Pomalidomide may stop the growth of blood vessels, stimulate the immune system, and kill cancer cells. Chemotherapy drugs, such as daunorubicin and cytarabine liposome, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Adding pomalidomide to chemotherapy treatment with daunorubicin and cytarabine liposome may be effective in improving some treatment outcomes in patients with newly diagnosed acute leukemia with myelodysplastic syndrome-related changes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish recommended phase 2 dose (RP2D) of pomalidomide after liposome-encapsulated daunorubicin-cytarabine (daunorubicin and cytarabine liposome) induction.

II. To compare the rate of overall complete response (CR)/complete response with incomplete hematologic recovery (CRi) with daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed acute myeloid leukemia (AML) with preexisting myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), or myeloproliferative neoplasm (MPN); therapy-related AML (t-AML); or AML with myelodysplasia-related changes (MRC) based on cytogenetics or morphologic dysplasia.

SECONDARY OBJECTIVES:

I. To evaluate and compare rates of CR (full hematologic recovery) between daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML or AML with MRC.

II. To evaluate and compare toxicities (including treatment-related mortality) of daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

III. To detect and compare the presence of minimal residual disease (MRD) by flow cytometry in those who achieve CR/CRi with daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

IV. To compare median event-free survival (EFS) of daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

V. To compare median overall survival (OS) of daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

VI. To compare median and 2-year disease-free survival (DFS) after CR/CRi with daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

VII. To compare rates of allogeneic stem cell transplant (SCT) after daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

EXPLORATORY OBJECTIVES:

I. To assess for molecular biomarkers, Aiolos expression, and immune correlates of response with daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

II. To assess for differences in MRD by molecular based platforms in daunorubicin and cytarabine liposome + pomalidomide versus daunorubicin and cytarabine liposome alone in newly diagnosed AML with preexisting MDS, CMML or MPN, t-AML, or AML with MRC based on cytogenetics or morphologic dysplasia.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A:

INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5 and then pomalidomide orally (PO) once daily (QD) beginning between days 21-30 for 14 days in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.

ARM B:

INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.

After completion of study treatment, patients are followed up for 30 days, then up to 5 years after the start of induction therapy or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of AML as defined by histologic, morphologic, or cytological evidence/confirmation of >= 20% blasts in bone marrow aspirate and/or biopsy
* Must meet criteria for t-AML or AML with MRC as defined by the 5th Edition of the World Health Organization (WHO) Classification of Myeloid Neoplasms or the International Consensus Classification (ICC) of Myeloid Neoplasms. Patients must meet one of the following criteria:

  * Therapy-related AML (AML derived from prior chemotherapy or radiation therapy)
  * AML originating from prior hematologic malignancy (MDS, CMML, or MPN)
  * AML with myelodysplasia-related cytogenetic abnormalities:

    * One of the following cytogenetic abnormalities:

      * Complex karyotype (3 or more unrelated chromosomal abnormalities in the absence of other class-defining recurrent genetic abnormalities as defined by WHO or ICC)
      * -7/del(7q)
      * Del(5q)/t(5q)/add(5q)
      * +8
      * i(17q)
      * -17/add(17p) or del(17p)
      * Del(20q)
      * -13/del(13q)
      * Del(11q)
      * Del(12p)/t(12p)/add(12p)
      * idicX(q13)
  * AML with myelodysplasia-related mutations: Must have a mutation in one of the following genes:

    * ASXL1
    * BCOR
    * EZH2
    * RUNX1
    * SF3B1
    * SRSF2
    * STAG2
    * U2AF1
    * ZRSR2
* No prior treatment for AML other than cytoreductive doses of hydroxyurea or leukapheresis
* Age >= 18 and =< 75 years on day of signing informed consent are eligible who are planned for intensive chemotherapy. Because no dosing or adverse event data are currently available on the use of pomalidomide in combination with daunorubicin and cytarabine liposome in patients < 18 years of age, children are excluded from this study. Patients > 75 years are not candidates for intensive chemotherapy with daunorubicin and cytarabine liposome
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Karnofsky >= 60%)
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN) unless due to leukemic infiltration, Gilbert's Syndrome, or hemolysis
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional ULN
* Creatinine >= 30 ml/min creatinine clearance by Cockcroft-gault
* Left ventricular ejection fraction (LVEF) >= 50%
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured with undetectable HCV viral load. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Females of childbearing potential (FCBP), defined as a female who: 1) has reached menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) must have a negative pregnancy test 72 hours prior to the start of study therapy. For FCBPs in Arm A, they must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients with Wilson's Disease or Copper-related metabolic disorders
* Absolute blast count > 30 x 10^9/L (cytoreduction with leukapheresis or hydroxyurea can be used to achieve absolute blast count < 30 x 10^9/L prior to day 1 of treatment)
* Cumulative daunorubicin lifetime exposure > 330 mg/m^2 and > 180 mg/m^2 with prior mediastinal radiation therapy
* Patients with known active central nervous system leukemia should be excluded from this clinical trial because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients receiving intrathecal chemotherapy prophylaxis should receive pomalidomide >= 3 days after administration
* Patients with uncontrolled intercurrent illness including, but not limited to, active and uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, and cardiac arrhythmia. Patients with infection under active treatment and controlled with antibiotics are eligible
* Known additional malignancy (with the exception of prior hematologic malignancies that have transformed to AML) that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical cancer or patients receiving maintenance treatments without active disease (for example, hormonal therapy for breast cancer or prostate cancer or other adjuvant chemotherapy approaches). Anti-cancer therapy as above should be discontinued > 72 hours prior to day 1 of treatment
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Receipt of prior allogeneic stem cell transplant
* Administration of any therapy for MDS, CMML, or MPN (conventional or unconventional) must be completed by 2 weeks prior to treatment with daunorubicin and cytarabine liposome. Use of strong CYP1A2 inhibitors should be avoided
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pomalidomide (e.g. lenalidomide, thalidomide) or daunorubicin and cytarabine liposome or their excipients
* Development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide, or similar drugs in the past
* Pregnant women are excluded from this study because pomalidomide is an immunomodulatory agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pomalidomide, breastfeeding should be discontinued if the mother is treated with pomalidomide. These potential risks may also apply to other agents used in this study. Women of childbearing potential must be willing to undergo pregnancy testing
* Any other medical condition that in the opinion of investigator would place patient at increased risk for toxicity during pomalidomide treatment (i.e. history of recurrent or serious thromboembolic events such as massive pulmonary embolism)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2026-04-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F Zeidner, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (11):
- United States (11):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - NYP/Weill Cornell Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant who was consented to the study declined to participate before being randomized to an arm.
Groups:
- Safety Run In DL1 (14 Days Pomalidomide): Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 and then pomalidomide PO QD beginning between days 21-30 for 14 days in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.
  Biospecimen Collection: Undergo collection of blood samples
  Bone Marrow Aspiration and Biopsy: Undergo bone marrow aspirate and biopsy
  Liposome-encapsulated Daunorubicin-Cytarabine: Given IV
  Pomalidomide: Given PO
- Safety Run In DL-1 (10 Days Pomalidomide): Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 and then pomalidomide PO QD beginning between days 21-30 for 10 days in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.
  Biospecimen Collection: Undergo collection of blood samples
  Bone Marrow Aspiration and Biopsy: Undergo bone marrow aspirate and biopsy
  Liposome-encapsulated Daunorubicin-Cytarabine: Given IV
  Pomalidomide: Given PO
- Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide): INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 and then pomalidomide PO QD beginning between days 21-30 for 14 days in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.
  Biospecimen Collection: Undergo collection of blood samples
  Bone Marrow Aspiration and Biopsy: Undergo bone marrow aspirate and biopsy
  Liposome-encapsulated Daunorubicin-Cytarabine: Given IV
  Pomalidomide: Given PO
- Arm B (Daunorubicin and Cytarabine Liposome): INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. Patients who do not respond, may receive a second cycle of liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 21 days for 2 cycles in the absence of disease progression and unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy and collection of blood samples throughout all phases of the trial.
  Biospecimen Collection: Undergo collection of blood samples
  Bone Marrow Aspiration and Biopsy: Undergo bone marrow aspirate and biopsy
  Liposome-encapsulated Daunorubicin-Cytarabine: Given IV
Period: Overall Study
Arm/Group | Safety Run In DL1 (14 Days Pomalidomide) | Safety Run In DL-1 (10 Days Pomalidomide) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) | Arm B (Daunorubicin and Cytarabine Liposome)
Started | 7 | 3 | 20 | 19
Completed | 6 | 3 | 16 | 18
Not Completed | 1 | 0 | 4 | 1
Not completed — Alternate Therapy prior to Day 21 | 1 | 0 | 1 | 1
Not completed — Clinical Instability | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run In DL1 (14 Days Pomalidomide) | Safety Run In DL-1 (10 Days Pomalidomide) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) | Arm B (Daunorubicin and Cytarabine Liposome) | Total
Number analyzed (Participants) | 6 | 3 | 16 | 18 | 43
Age, Continuous [Median (Full Range); unit: years] | 68.5 [23 to 73] | 66 [62 to 69] | 63 [49 to 74] | 63 [34 to 74] | 63 [23 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 9 | 10 | 26
  Male | 1 | 1 | 7 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 3 | 15 | 18 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 1 | 4
  White | 5 | 3 | 12 | 15 | 35
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 16 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response (CR)/Complete Response With Incomplete Hematologic Recovery (CRi)
Time Frame: Up to 2 years
Population: This outcome measure was not reported on for the safety run-in phase
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run In DL1 (14 Days Pomalidomide) | Safety Run In DL-1 (10 Days Pomalidomide) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) | Arm B (Daunorubicin and Cytarabine Liposome)
Number analyzed (Participants) | 0 | 0 | 16 | 18
Participants |  |  | 9 | 13

2. Secondary Outcome: CR With Full Hematologic Recovery (Absolute Neutrophil Count > 1 x 10^9/L and Platelets > 100 x 10^9/L)
Description: Will be assessed and compared with both arms A and B.
Time Frame: Up to 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5.0 and compared descriptively between Arms A and B. Serious adverse events are denoted by "[SAE]".
Time Frame: Up to 30 days after last dose, up to 2 years
Measure: Number; unit: participants
Arm/Group | Safety Run In DL1 (14 Days Pomalidomide) | Safety Run In DL-1 (10 Days Pomalidomide) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) | Arm B (Daunorubicin and Cytarabine Liposome)
Number analyzed (Participants) | 7 | 3 | 20 | 19
participants
  Alanine Aminotransferase Increased | 4 | 2 | 8 | 8
  Aspartate Aminotransferase Increased | 6 | 2 | 8 | 8
  Abdominal Distension | 0 | 0 | 1 | 0
  Activated Partial Thromboplastin Time Prolonged | 0 | 0 | 2 | 0
  Acute Kidney Injury | 0 | 0 | 1 | 0
  Alkaline Phosphatase Increased | 4 | 2 | 7 | 4
  Alkalosis | 1 | 0 | 0 | 0
  Allergic Reaction | 1 | 0 | 0 | 0
  Alopecia | 0 | 0 | 1 | 0
  Anal fissure | 0 | 0 | 1 | 0
  Anal Fistula | 1 | 0 | 0 | 1
  Atrial Flutter | 0 | 0 | 1 | 0
  Back Pain | 0 | 0 | 2 | 1
  Bacteremia | 1 | 1 | 4 | 5
  Bloating | 0 | 0 | 2 | 1
  Blood Bicarbonate Decreased | 0 | 0 | 1 | 0
  Blood Bilirubin Increased | 4 | 2 | 6 | 3
  Blood/Lymph - Other - D Dimer increased | 0 | 0 | 1 | 0
  Blood/Lymph - Other - Increased Fibrinogen | 0 | 0 | 1 | 1
  Blood/Lymph - Other - PT increased | 0 | 0 | 1 | 0
  Blood/Lymph - Other - febrile non-hemolytic transfusion reaction (FNHTR) | 0 | 0 | 1 | 0
  Blood/Lymph - Other - petechiae | 0 | 0 | 0 | 2
  Burred Vision | 0 | 0 | 0 | 3
  Bone Pain | 0 | 0 | 2 | 1
  Bruising | 1 | 0 | 1 | 0
  Cardiac Troponin I Increased | 1 | 0 | 0 | 0
  Catheter Related Infection | 0 | 0 | 1 | 0
  Chest Wall Pain | 0 | 0 | 2 | 0
  Chills | 0 | 1 | 4 | 2
  Chronic Kidney Disease | 0 | 0 | 1 | 0
  Confusion | 0 | 1 | 1 | 1
  Constipation | 4 | 0 | 12 | 10
  Cough | 0 | 3 | 7 | 5
  Creatinine Increased | 3 | 0 | 4 | 3
  Cytokine Release Syndrome | 0 | 0 | 1 | 0
  Disseminated Intravascular Coagulation | 0 | 0 | 0 | 2
  Dehydration | 0 | 0 | 0 | 2
  Delirium | 2 | 0 | 0 | 0
  Delusions | 0 | 1 | 0 | 0
  Depression | 0 | 1 | 0 | 1
  Diarrhea | 2 | 1 | 6 | 4
  Dizziness | 1 | 1 | 4 | 4
  Dry Mouth | 0 | 1 | 2 | 1
  Dysgeusia | 0 | 1 | 3 | 2
  Dyspepsia | 1 | 0 | 0 | 1
  Dysphagia | 0 | 0 | 0 | 1
  Dyspnea | 2 | 1 | 9 | 1
  EKG QT Corrected Interval Prolong | 0 | 0 | 1 | 0
  Ear and Labyrinth - Other - Serous otitis media | 0 | 0 | 0 | 1
  Ear Pain | 0 | 0 | 1 | 0
  Edema Face | 0 | 0 | 1 | 1
  Edema Limbs | 2 | 2 | 8 | 6
  Elevated Lactate Dehydrogenase (LDH) | 1 | 1 | 3 | 4
  Eosinophilia | 2 | 0 | 0 | 0
  Epistaxis | 1 | 2 | 5 | 6
  Esophageal Hemorrhage | 0 | 0 | 0 | 1
  Extrapyramidal Disorder | 0 | 0 | 0 | 1
  Fall | 0 | 0 | 2 | 1
  Fatigue | 3 | 3 | 8 | 6
  Febrile Neutropenia | 2 | 1 | 8 | 4
  Fever | 1 | 1 | 4 | 4
  Fibrinogen Decreased | 0 | 1 | 1 | 0
  Flatulence | 0 | 0 | 2 | 2
  Floaters | 0 | 0 | 0 | 1
  Flushing | 0 | 0 | 0 | 1
  Folliculitis | 0 | 1 | 0 | 0
  Gamma-Glutamyl Transferase (GGT) Increased | 0 | 0 | 1 | 0
  GI disorders - Other, specify - Black lesion on tongue | 0 | 0 | 0 | 1
  GI disorders - Other, specify - Bright red blood per rectum | 0 | 0 | 1 | 0
  GI disorders - Other, specify - Diverticulitis | 0 | 0 | 1 | 0
  GI disorders - Other, specify - Gastrointestinal bleeding | 0 | 1 | 0 | 0
  GI disorders - Other, specify - Genitourinary bleeding | 0 | 0 | 0 | 1
  GI disorders - Other, specify - Gum Bleeding | 0 | 0 | 1 | 1
  GI disorders - Other, specify - Lip lesion | 0 | 0 | 0 | 1
  GI disorders - Other, specify - Lower GI hemmorrage | 0 | 0 | 1 | 0
  GI disorders - Other, specify - Melena | 0 | 0 | 1 | 1
  GI disorders - Other, specify - Rectal bleeding | 0 | 0 | 1 | 0
  GI disorders - Other, specify - Wet Purpura | 0 | 0 | 1 | 0
  GI disorders - Other, specify - hematochezia | 0 | 0 | 1 | 0
  Gastroesophageal reflux disease | 0 | 0 | 2 | 0
  Gastrointestinal Pain | 1 | 0 | 1 | 0
  Generalized Edema | 2 | 0 | 2 | 0
  Generalized Muscle Weakness | 0 | 0 | 3 | 1
  Genital Edema | 0 | 0 | 0 | 1
  Headache | 2 | 2 | 5 | 7
  Hearing Impaired | 0 | 0 | 0 | 1
  Heart Failure | 0 | 0 | 1 | 0
  Hematoma | 0 | 0 | 1 | 1
  Hematuria | 2 | 1 | 2 | 2
  Hemorrhoidal Hemorrhage | 0 | 1 | 0 | 0
  Hemorrhoids | 1 | 0 | 0 | 1
  Hoarseness | 0 | 0 | 0 | 1
  Hypercalcemia | 1 | 0 | 0 | 1
  Hyperglycemia | 1 | 0 | 6 | 6
  Hyperhidrosis | 1 | 0 | 0 | 0
  Hyperkalemia | 2 | 1 | 2 | 1
  Hypermagnesemia | 0 | 0 | 1 | 2
  Hypernatremia | 2 | 0 | 1 | 1
  Hyperphosphatemia | 1 | 1 | 2 | 5
  Hypertension | 0 | 1 | 5 | 6
  Hyperuricemia | 0 | 0 | 0 | 1
  Hypoalbuminemia | 7 | 3 | 12 | 14
  Hypocalcemia | 3 | 1 | 8 | 9
  Hypokalemia | 6 | 2 | 10 | 11
  Hypomagnesemia | 2 | 0 | 4 | 3
  Hyponatremia | 4 | 2 | 7 | 10
  Hypophosphatemia | 3 | 2 | 5 | 4
  Hypotension | 0 | 1 | 3 | 3
  Hypoxia | 0 | 0 | 3 | 2
  International Normalized Ratio (INR) Increased | 0 | 1 | 3 | 1
  Infections & infestations - Other - Pediculosis captis | 0 | 0 | 1 | 0
  Infections & infestations - Other - Sars-COV-2 | 0 | 0 | 1 | 0
  Infections & infestations - Other - Sepsis | 1 | 0 | 1 | 0
  Infusion Related Reaction | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - Acute RLE DVT | 0 | 0 | 1 | 0
  Injury/poison/procedure - Other - Acute RUE VTE (superficial and deep) | 0 | 0 | 1 | 0
  Injury/poison/procedure - Other - Central line incision site erythema | 0 | 0 | 1 | 0
  Injury/poison/procedure - Other - L maxillary anterior, medial, posterior wall fracture | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - L nasal dorsum laceration | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - Left lateral orbital wall fracture | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - R orbital roof/lateral orbital wall fracture | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - Septal fracture | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - bilateral nasal bone fracture | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - left frontal bone fracture | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - left inferior orbital wall fracture | 0 | 0 | 0 | 1
  Injury/poison/procedure - Other - left supraorbital laceration | 0 | 0 | 0 | 1
  Insomnia | 3 | 1 | 5 | 5
  Investigations - Other, specify - Hyperfibrinogenemia | 0 | 0 | 1 | 0
  Investigations - Other, specify - Increased Fibrinogen | 0 | 0 | 1 | 0
  Investigations - Other, specify - increased chloride | 0 | 0 | 1 | 0
  Localized Edema | 0 | 1 | 2 | 0
  Lung Infection | 0 | 0 | 2 | 5
  Lymph Node Pain | 1 | 0 | 0 | 0
  Lymphocyte Count Decreased | 5 | 2 | 12 | 13
  Lymphocyte Count Increased | 0 | 0 | 1 | 0
  Mucositis Oral | 3 | 1 | 9 | 5
  Muscle Cramp | 0 | 0 | 0 | 1
  Muscle Weakness Upper Limb | 0 | 0 | 1 | 0
  Musculoskel/connect tissue -Other - Blanchable tissue (Buttocks) | 0 | 0 | 0 | 1
  Musculoskel/connect tissue -Other - Deep tissue injury (buttocks) | 0 | 0 | 0 | 1
  Musculoskel/connect tissue -Other - Pain in LLE | 1 | 0 | 0 | 0
  Musculoskel/connect tissue -Other - vastus lateralis muscle strain | 0 | 0 | 0 | 1
  Myalgia | 0 | 0 | 0 | 2
  Nasal Congestion | 3 | 0 | 1 | 6
  Nausea | 6 | 2 | 8 | 8
  Neck Pain | 0 | 0 | 3 | 1
  Nervous system - Other - Anomia | 0 | 1 | 0 | 0
  Nervous system - Other - Rigors | 0 | 0 | 0 | 1
  Neutrophil Count Decreased | 7 | 2 | 11 | 11
  Non-cardiac Chest Pain | 0 | 1 | 1 | 1
  Oral Hemorrhage | 0 | 1 | 1 | 1
  Oral Pain | 2 | 1 | 1 | 2
  Pain | 0 | 1 | 5 | 6
  Pain in Extremity | 0 | 1 | 1 | 4
  Papulopustular Rash | 0 | 1 | 1 | 0
  Paresthesia | 1 | 0 | 0 | 0
  Pericardial Effusion | 0 | 0 | 2 | 0
  Periodontal Disease | 0 | 0 | 0 | 1
  Peripheral Motor Neuropathy | 1 | 0 | 0 | 0
  Peripheral Sensory Neuropathy | 0 | 0 | 0 | 2
  Pharyngitis | 0 | 0 | 1 | 0
  Platelet Count Decreased | 7 | 3 | 16 | 12
  Pleural Effusion | 0 | 0 | 4 | 5
  Pleuritic Pain | 0 | 0 | 0 | 1
  Presyncope | 0 | 0 | 0 | 1
  Proctitis | 0 | 0 | 2 | 0
  Productive Cough | 1 | 0 | 0 | 1
  Proteinuria | 1 | 2 | 1 | 1
  Pruritus | 1 | 1 | 4 | 6
  Pulmonary Edema | 1 | 0 | 3 | 0
  Pulmonary Hypertension | 0 | 0 | 0 | 1
  Purpura | 1 | 0 | 0 | 0
  Rash Maculo-papular | 4 | 1 | 8 | 8
  Rectal Hemorrhage | 0 | 0 | 0 | 1
  Rectal Pain | 0 | 0 | 0 | 3
  Resp, thoracic & mediast - Other - Hemoptysis | 0 | 0 | 0 | 1
  Resp, thoracic & mediast - Other - Nasal dryness | 0 | 0 | 1 | 0
  Resp, thoracic & mediast - Other - Nasal irritation | 0 | 0 | 0 | 1
  Respiratory Failure | 0 | 0 | 1 | 0
  Restlessness | 1 | 0 | 0 | 0
  Retinal Tear | 0 | 0 | 0 | 1
  Rhinorrhea | 1 | 0 | 0 | 1
  Scrotal Pain | 2 | 0 | 0 | 0
  Sepsis | 0 | 0 | 1 | 0
  Sinus Bradycardia | 0 | 1 | 3 | 0
  Sinus Tachycardia | 0 | 0 | 2 | 0
  Skin & subcutaneous tissue -Other - Actinic Keratosis Reaction | 0 | 1 | 0 | 0
  Skin & subcutaneous tissue -Other - Back Lesion | 0 | 0 | 1 | 0
  Skin & subcutaneous tissue -Other - Erythema around line insertion | 0 | 0 | 1 | 0
  Skin & subcutaneous tissue -Other - L Ankle lesion | 0 | 0 | 1 | 0
  Skin & subcutaneous tissue -Other - L skin lesion (Wrist) | 0 | 0 | 1 | 0
  Skin & subcutaneous tissue -Other - Petechial rash | 0 | 0 | 1 | 0
  Skin & subcutaneous tissue -Other - Purulence at site of prior picc line | 0 | 0 | 1 | 0
  Skin & subcutaneous tissue -Other - R leg nodules | 0 | 0 | 0 | 1
  Skin & subcutaneous tissue -Other - R leg subcu nodules | 0 | 0 | 0 | 1
  Skin & subcutaneous tissue -Other - Right neck rash | 0 | 0 | 0 | 1
  Skin & subcutaneous tissue -Other - nodule | 0 | 0 | 0 | 1
  Skin Infection | 0 | 1 | 2 | 3
  Soft Tissue Infection | 0 | 0 | 0 | 1
  Sore Throat | 1 | 0 | 2 | 1
  Supraventricular Tachycardia | 0 | 0 | 0 | 1
  Thromboembolic Event | 1 | 0 | 0 | 1
  Thrush | 0 | 0 | 2 | 2
  Tremor | 1 | 0 | 1 | 0
  Typhlitis | 0 | 0 | 3 | 0
  Upper Gastrointestinal Hemorrhage | 0 | 0 | 1 | 0
  Upper Respiratory Infection | 0 | 0 | 1 | 0
  Urinary Frequency | 0 | 1 | 1 | 1
  Urinary Incontinence | 1 | 0 | 0 | 1
  Urinary Retention | 0 | 0 | 2 | 0
  Urinary Urgency | 0 | 0 | 0 | 2
  Vaginal Hemorrhage | 0 | 0 | 0 | 1
  Vaginal Pain | 0 | 0 | 0 | 1
  Vascular Access Complication | 2 | 0 | 8 | 9
  Ventricular Arrhythmia | 0 | 0 | 0 | 1
  Vomiting | 2 | 1 | 6 | 4
  Weight Gain | 1 | 1 | 1 | 1
  Weight Loss | 0 | 1 | 2 | 0
  Wheezing | 0 | 1 | 0 | 0
  White Blood Cell Decreased | 5 | 3 | 16 | 14
  [SAE] Alanine Aminotransferase (ALT) Increased | 1 | 1 | 2 | 1
  [SAE] Acute Respiratory Distress Syndrome (ARDS) | 0 | 0 | 1 | 0
  [SAE] Aspartate Aminotransferase (AST) Increased | 2 | 1 | 2 | 3
  [SAE] Abdominal Pain | 0 | 0 | 1 | 0
  [SAE] Activated Partial Thromboplastin Time (PTT) Prolonged | 0 | 0 | 1 | 0
  [SAE] Acute Kidney Injury | 1 | 0 | 1 | 0
  [SAE] Alkaline phosphatase increased | 0 | 1 | 2 | 0
  [SAE] Anemia | 7 | 3 | 13 | 11
  [SAE] Anorexia | 1 | 0 | 0 | 0
  [SAE] Anxiety | 0 | 0 | 0 | 1
  [SAE] Atrial Fibrillation | 0 | 0 | 2 | 0
  [SAE] Atrial Flutter | 0 | 0 | 1 | 0
  [SAE] Blood Bilirubin Increased | 0 | 1 | 3 | 0
  [SAE] Cardiac Arrest | 0 | 0 | 1 | 0
  [SAE] Catheter Related Infection | 0 | 0 | 1 | 0
  [SAE] Creatinine Incrased | 1 | 0 | 0 | 0
  [SAE] Delirium | 2 | 0 | 0 | 0
  [SAE] Disease Progression | 1 | 0 | 2 | 0
  [SAE] Dyspnea | 1 | 0 | 4 | 1
  [SAE] EKG QT corrected interval prolong | 1 | 0 | 0 | 0
  [SAE] Eosinophilia | 1 | 0 | 0 | 0
  [SAE] Epistaxis | 0 | 0 | 0 | 2
  [SAE] Eye disorders - Other, specify - Right eye vision lost | 0 | 0 | 1 | 0
  [SAE] Fall | 0 | 0 | 0 | 1
  [SAE] Fatigue | 1 | 0 | 0 | 0
  [SAE] Febrile Neutropenia | 5 | 3 | 14 | 16
  [SAE] GI disorders - Other, specify - Diverticulitis | 0 | 0 | 1 | 0
  [SAE] GI disorders - Other, specify - melena | 0 | 0 | 1 | 0
  [SAE] Heart Failure | 0 | 0 | 1 | 0
  [SAE] Hematuria | 0 | 0 | 1 | 0
  [SAE] Hyperkalemia | 1 | 0 | 0 | 0
  [SAE] Hypertension | 0 | 0 | 5 | 4
  [SAE] Hypoalbuminemia | 1 | 1 | 3 | 2
  [SAE] Hypocalcemia | 1 | 0 | 0 | 0
  [SAE] Hypokalemia | 1 | 2 | 3 | 4
  [SAE] Hypotension | 0 | 0 | 2 | 1
  [SAE] Hypoxia | 0 | 0 | 8 | 2
  [SAE] Infections & infestations - Other - Sepsis | 2 | 0 | 4 | 2
  [SAE] Lung Infection | 1 | 2 | 3 | 4
  [SAE] Lymphocyte Count Decreased | 4 | 2 | 11 | 12
  [SAE] Lymphocyte Count Increased | 0 | 0 | 1 | 0
  [SAE] Nausea | 1 | 0 | 0 | 0
  [SAE] Neutrophil Count Decreased | 7 | 2 | 12 | 11
  [SAE] Platelet Count Decreased | 7 | 3 | 17 | 13
  [SAE] Pleural Effusion | 0 | 1 | 0 | 2
  [SAE] Pulmonary Edema | 0 | 0 | 3 | 2
  [SAE] Rash Maculo-papular | 0 | 0 | 0 | 1
  [SAE] Rectal Pain | 0 | 0 | 0 | 1
  [SAE] Renal Calculi | 0 | 0 | 1 | 0
  [SAE] Respiratory Failure | 0 | 0 | 1 | 0
  [SAE] Seizure | 0 | 0 | 1 | 0
  [SAE] Sepsis | 1 | 0 | 2 | 0
  [SAE] Sinus Bradycardia | 0 | 0 | 1 | 0
  [SAE] Sinusitis | 0 | 0 | 1 | 0
  [SAE] Skin Infection | 0 | 1 | 1 | 2
  [SAE] Soft Tissue Infection | 0 | 0 | 0 | 1
  [SAE] Supraventricular Tachycardia | 0 | 0 | 0 | 1
  [SAE] Syncope | 0 | 0 | 0 | 1
  [SAE] Typhlitis | 0 | 0 | 3 | 0
  [SAE] Upper Gastrointestinal Hemorrhage | 0 | 0 | 2 | 0
  [SAE] Urinary Retention | 0 | 0 | 1 | 0
  [SAE] Vascular Access Complication | 0 | 0 | 2 | 1
  [SAE] Vomiting | 1 | 0 | 0 | 0
  [SAE] White Blood Cell Decreased | 6 | 3 | 16 | 15

4. Secondary Outcome: Complete Response (CR) Without Minimal Residual Disease (MRD)
Description: Will assess CR without MRD by flow cytometry via Hematologics, Inc. compare descriptively between Arms A and B.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Event-free Survival
Description: Will be compared between Arms A and B.
Time Frame: From day 1 of liposome-encapsulated daunorubicin-cytarabine until no response is achieved, relapse or death, will be assessed for up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Disease-free Survival (DFS)
Description: Will be compared between Arms A and B.
Time Frame: From CR/CRi until relapse or death, assessed at 2 years
Population: This outcome measure was not reported on for the safety run-in phase
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety Run In DL1 (14 Days Pomalidomide) | Safety Run In DL-1 (10 Days Pomalidomide) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) | Arm B (Daunorubicin and Cytarabine Liposome)
Number analyzed (Participants) | 0 | 0 | 16 | 18
months |  |  | 8.18 [6.28 to NA] — Upper confidence interval is not available due to insufficient number of events | NA [NA to NA] — Median DFS is not available due to insufficient number of events

7. Secondary Outcome: Disease-free Survival
Description: Will be compared between Arms A and B.
Time Frame: From CR/CRi until relapse or death, assessed up to 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Overall Survival (OS)
Description: Will be compared between Arms A and B.
Time Frame: From randomization until death or last follow-up, assessed up to 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Rate of Allogeneic Stem Cell Transplantation
Description: Will be compared between Arms A and B.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose, up to 2 years
Arm/Group | Safety Run In DL1 (14 Days Pomalidomide) | Safety Run In DL-1 (10 Days Pomalidomide) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) | Arm B (Daunorubicin and Cytarabine Liposome)
All-Cause Mortality (participants affected / at risk) | 3/7 | 2/3 | 11/20 | 7/19
Serious Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 19/20 | 19/19
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 20/20 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run In DL1 (14 Days Pomalidomide) (N=7) | Safety Run In DL-1 (10 Days Pomalidomide) (N=3) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) (N=20) | Arm B (Daunorubicin and Cytarabine Liposome) (N=19)
Alanine Aminotransferase Increased (Investigations) | 1 (3) | 1 (3) | 2 (3) | 1 (2)
Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 2 (4) | 1 (3) | 2 (10) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (60) | 3 (21) | 13 (76) | 11 (49)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (8) | 3 (12) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 4 (5) | 1 (1)
EKG QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Eye disorders - Other, specify - Right eye vision lost (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (12) | 3 (6) | 14 (34) | 16 (27)
GI disorders - Other, specify - melena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI disorders - Other, specify - Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 5 (12) | 4 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (4) | 1 (3) | 3 (7) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (6) | 3 (9) | 4 (10)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (10) | 2 (3)
Infections & infestations - Other - Sepsis (Infections and infestations) | 2 (5) | 0 (0) | 4 (5) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1) | 2 (3) | 3 (11) | 4 (12)
Lymphocyte Count Decreased (Investigations) | 4 (29) | 2 (10) | 11 (87) | 12 (64)
Lymphocyte Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 7 (31) | 2 (19) | 12 (54) | 11 (45)
Platelet count decreased (Investigations) | 7 (110) | 3 (35) | 17 (122) | 13 (79)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (4) | 2 (3)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White Blood Cell Decreased (Investigations) | 6 (31) | 3 (32) | 16 (86) | 15 (73)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run In DL1 (14 Days Pomalidomide) (N=7) | Safety Run In DL-1 (10 Days Pomalidomide) (N=3) | Arm A (Daunorubicin and Cytarabine Liposome, Pomalidomide) (N=20) | Arm B (Daunorubicin and Cytarabine Liposome) (N=19)
Alanine Aminotransferase Increased (Investigations) | 4 (17) | 2 (10) | 8 (24) | 8 (27)
Aspartate Aminotransferase Increased (Investigations) | 6 (25) | 2 (16) | 8 (34) | 8 (36)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 6 (12) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 4 (10) | 2 (15) | 7 (18) | 4 (9)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 7 (106) | 3 (32) | 13 (116) | 11 (104)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 4 (5) | 5 (8)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (3) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (3)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1) | 4 (7) | 5 (5)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood Bicarbonate Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 4 (17) | 2 (13) | 6 (31) | 3 (4)
Blood/Lymph - Other - D Dimer increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood/Lymph - Other - Increased Fibrinogen (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Blood/Lymph - Other - Prothrombin Time increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood/Lymph - Other - febrile non-hemolytic transfusion reaction (FNHTR) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood/Lymph - Other - petechiae (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Cardiac Troponin I Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 4 (9) | 2 (2)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (7) | 0 (0) | 12 (21) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (7) | 7 (11) | 5 (5)
Creatinine Increased (Investigations) | 3 (16) | 0 (0) | 4 (4) | 3 (5)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated Intravascular Coagulation (DIC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Delirium (Psychiatric disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Delusions (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (12) | 4 (5)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (9)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (4) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 1 (3) | 9 (19) | 1 (1)
EKG QT corrected interval prolong (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear and Labyrinth - Other - Serous otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Edema Face (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Edema limbs (General disorders) | 2 (3) | 2 (2) | 8 (19) | 6 (12)
Elevated Lactate Dehydrogenase (Investigations) | 1 (3) | 1 (2) | 3 (7) | 4 (7)
Eosinophilia (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 5 (7) | 6 (9)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Fatigue (General disorders) | 3 (11) | 3 (6) | 8 (19) | 6 (6)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 8 (15) | 4 (5)
Fever (General disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (4)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gamma-Glutamyl Transferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI disorders - Other, specify - Black lesion on tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI disorders - Other, specify - Bright red blood per rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
GI disorders - Other, specify - Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI disorders - Other, specify - Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
GI disorders - Other, specify - Genitourinary bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI disorders - Other, specify - Gum Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GI disorders - Other, specify - Lip lesion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI disorders - Other, specify - Lower GI hemmorrage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
GI disorders - Other, specify - Melena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
GI disorders - Other, specify - Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI disorders - Other, specify - Wet Purpura (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI disorders - Other, specify - hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (8) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Generalized Edema (General disorders) | 2 (5) | 0 (0) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (7) | 1 (1)
Genital Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 2 (4) | 5 (9) | 7 (15)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (2)
Hoarsenes (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 6 (19) | 6 (21)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 1 (4) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 5 (12) | 6 (10)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (49) | 3 (22) | 12 (72) | 14 (78)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (14) | 1 (7) | 8 (22) | 9 (26)
Hypokalemia (Metabolism and nutrition disorders) | 6 (31) | 2 (20) | 10 (68) | 11 (39)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 4 (5) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (17) | 2 (18) | 7 (23) | 10 (23)
Hypophospatemia (Metabolism and nutrition disorders) | 3 (10) | 2 (4) | 5 (8) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 3 (4) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
International Normalized Ratio (INR) Increased (Investigations) | 0 (0) | 1 (2) | 3 (4) | 1 (1)
Infections & infestations - Other - Pediculosis captis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections & infestations - Other - Sars-COV-2 (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infections & infestations - Other - Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury/poison/procedure - Other - Acute RLE DVT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury/poison/procedure - Other - Acute RUE VTE (superficial and deep) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injury/poison/procedure - Other - Central line incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injury/poison/procedure - Other - L maxillary anterior, medial, posterior wall fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injury/poison/procedure - Other - L nasal dorsum laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injury/poison/procedure - Other - Left lateral orbital wall fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injury/poison/procedure - Other - R orbital roof/lateral orbital wall fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injury/poison/procedure - Other - Septal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injury/poison/procedure - Other - bilateral nasal bone fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injury/poison/procedure - Other - left frontal bone fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injury/poison/procedure - Other - left inferior orbital wall fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injury/poison/procedure - Other - left supraorbital laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 3 (6) | 1 (2) | 5 (13) | 5 (7)
Investigations - Other, specify - Hyperfibrinogenemia (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Investigations - Other, specify - Increased Fibrinogen (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Investigations - Other, specify - increased chloride (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (6) | 2 (2) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (5) | 5 (7)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (56) | 2 (31) | 12 (114) | 13 (127)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (6) | 1 (2) | 9 (14) | 5 (8)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskel/connect tissue -Other - Blanchable tissue (Buttocks) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskel/connect tissue -Other - Deep tissue injury (buttocks) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskel/connect tissue -Other - Pain in LLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskel/connect tissue -Other - vastus lateralis muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 1 (2) | 6 (10)
Nausea (Gastrointestinal disorders) | 6 (9) | 2 (3) | 8 (11) | 8 (17)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Nervous system - Other - Anomia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nervous system - Other - Rigors (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 7 (26) | 2 (21) | 11 (47) | 11 (43)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (3)
Oral Pain (Gastrointestinal disorders) | 2 (3) | 1 (2) | 1 (2) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 5 (10) | 6 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (7)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 7 (113) | 3 (35) | 16 (106) | 12 (81)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (7) | 5 (5)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (2) | 2 (5) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 4 (6) | 6 (8)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (13) | 1 (2) | 8 (18) | 8 (16)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Resp, thoracic & mediast - Other - Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Resp, thoracic & mediast - Other - Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Resp, thoracic & mediast - Other - Nasal irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Retinal Tear (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Skin & subcutaneous tissue -Other - Actinic Keratosis Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin & subcutaneous tissue -Other - Back Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin & subcutaneous tissue -Other - Erythema around line insertion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin & subcutaneous tissue -Other - L Ankle lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin & subcutaneous tissue -Other - L skin lesion (Wrist) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin & subcutaneous tissue -Other - Petechial rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin & subcutaneous tissue -Other - Purulence at site of prior picc line (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin & subcutaneous tissue -Other - R leg nodules (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin & subcutaneous tissue -Other - R leg subcu nodules (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin & subcutaneous tissue -Other - Right neck rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin & subcutaneous tissue -Other - nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 8 (11) | 9 (13)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 6 (7) | 4 (6)
Weight gain (Investigations) | 1 (1) | 1 (3) | 1 (4) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 5 (38) | 3 (32) | 16 (84) | 14 (84)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT04802161/Prot_SAP_000.pdf
  • Informed Consent Form: P10434_A16ScreeningConsent(Untracked).pdf (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT04802161/ICF_001.pdf
  • Informed Consent Form: P10434_A16Consent(Untracked).pdf (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT04802161/ICF_002.pdf